CLINICAL TRIAL: NCT05306925
Title: An Exploratory Study of Arginine Supplementation and the Postoperative Immune REsponse (ASPIRE)
Brief Title: An Exploratory Study of Arginine Supplementation and the Postoperative Immune REsponse
Acronym: ASPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UoL001648
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Preterm; Surgery; Nutritional Deficiency; Immune System and Related Disorders
Keywords: Neonate; Arginine; Postoperative; Immune function; Nutrition
MeSH Terms: conditions — Premature Birth; Malnutrition | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: There will be parallel assignment of supplemented parenteral nutrition (PN) and standard parenteral nutrition dependent upon stock availability of intervention PN.
Masking Description: This is not blinded or randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard parenteral nutrition (No Intervention): These infants will form the control group and will receive standard parenteral nutrition. They will be sub-stratified into gestational brackets - preterm (born <30 weeks) and term/near term.
- Arginine supplementation (combined) (Experimental): These infants will form an intervention group and will receive parenteral nutrition with additional arginine (up to 18% of amino acid make-up) for up to 14 days post-op and oral arginine supplementation up to 30 days post-op. They will be sub-stratified into gestational brackets - preterm (born <30 weeks) and term/near term.
  Interventions: Dietary Supplement: Arginine
- Arginine supplementation (oral only) (Experimental): These infants will form an intervention group and will receive standard parenteral nutrition and oral arginine supplementation up to 30 days post-op. They will be sub-stratified into gestational brackets - preterm (born <30 weeks) and term/near term.
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — The intervention infants will receive either parenteral nutrition which contains additional arginine (up to 18% arginine content) or a separate arginine infusion to provide up to 18% arginine. This is in comparison to standard parenteral nutrition which has an arginine content of 6.3%.
  Arms: Arginine supplementation (combined); Arginine supplementation (oral only)

SUMMARY:
ASPIRE is a nutrition study focusing on the effect of arginine supplementation on immune function in postoperative infants.

The investigators will explore the effect of current intravenous feeding (parenteral nutrition (PN)) formulations and oral arginine supplementation on blood arginine levels and the genes that are involved in body nutrition and fighting infection in babies who have had major bowel surgery or been diagnosed with necrotising enterocolitis. The investigators will undertake an exploratory physiological study across two sites under which are part of a single neonatal partnership. 48 infants will be recruited; 24 preterm infants and 24 term/near term infants. 16 of these infants (8 preterm and 8 term/near term) will be supplemented with arginine in both oral and parenteral form, 16 infants will receive arginine supplementation in oral form alone and 16 infants will receive standard nutrition with no arginine supplement. The investigators will record nutritional intake and routine biochemical testing data (which includes amino acid levels) collected over the first 30 days post surgery or post NEC diagnosis. The investigators will take blood for analysis at prespecified intervals for RNA sequencing, ammonia and metabolomics. RNA sequencing findings will allow the investigators to describe the effect of arginine on gene activity in postoperative infants

The investigators hypothesise that arginine supplementation will result in changes in gene expression that are consistent with changes in T-cell function and associated inflammatory pathways.

DETAILED DESCRIPTION:
Title:

Arginine Supplementation and the Postoperative Immune REsponse (ASPIRE) in neonates

Population:

Preterm infants <30 weeks gestation requiring a laparotomy/major bowel surgery or diagnosed with necrotising enterocolitis (Modified Bell's Stage II or higher) before discharge before discharge ; Term and near term infants (born >35 weeks gestation) requiring a laparotomy/major bowel surgery in the first 3 days of life (gastroschisis; major bowel atresias expected to require at least 7 days PN).

Number of infants:

48 infants (completing the study) will be recruited over approximately 24-36 months: 24 in the preterm group and 24 in the term group.

Number of sites:

Two sites - Alder Hey Children's Hospital (AHCH) and Liverpool Women's Hospital (LWH) under the umbrella of the Neonatal Partnership. Eligible infants will undergo surgery at AHCH and will receive early postoperative care at either AHCH or LWH

Study duration:

Informed consent will take place preoperatively where possible, or within 5 days of surgery or NEC diagnosis. In the term group, antenatal recruitment will be attempted. The first study related blood sample will be taken as soon as possible postoperatively following consent with the last sample taken on day 30 post-operatively. Other study assessments reflect those routinely performed in preterm infants receiving parenteral nutrition (PN).

Study intervention:

All infants will receive standard clinical treatment. 8 preterm and 8 term infants will receive PN as determined by local clinical guidelines (6.3 or 8.4% arginine content). 8 term infants and 8 preterm infants will receive PN as determined by local clinical guidelines (6.3 or 8.4% arginine content) and enteral arginine supplementation. Enteral L-arginine will start with the first enteral feedings: starting 0.75mmol/kg/day, doubled to 1.5mmol/kg (261mg/kg/day) when reaching 40% of enteral feeds. 8 preterm and 8 term infants will receive PN with an additional arginine supplement and oral supplementation. PN supplementation will aim to achieve up to 18% arginine intake (allocated according to intervention PN stock availability) and will be titrated against oral supplementation during the transition to enteral feeds.

Primary objective:

To examine the changes in gene expression present in arginine supplemented infants between day 3 and day 10 post-operatively. Thus will be done via illumina RNA sequencing and statistical pathway analysis. The changes in gene expression will be compared with those seen between day 3 and day 10 in unsupplemented preterm and term infants. The genes of interest are those involved in immune function and inflammatory pathways.

Secondary objectives:

1. To explore other biological pathways i) known to be involved in the pathogenesis of necrotising enterocolitis ii) involved in arginine metabolism iii) that are related to the insulin-IGF-I axis
2. To determine the changes in metabolomic profiles of these infants during the first 30 days postoperatively.
3. Growth and body composition data during study period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born <30 weeks gestation requiring laparotomy/major bowel surgery or diagnosed with necrotising enterocolitis (Modified Bell's Stage II or higher) before discharge
* Term and near term infants (born>35 weeks gestation) requiring laparotomy/major bowel surgery in the first 3 days of life (gastroschisis; major bowel atresias expected to require at least 7 days of PN)

Exclusion Criteria:

* Infants who are unlikely to survive because of poor immediate postoperative condition
* Infants known (or suspected to have) a diagnosis of inborn error of metabolism or serious liver dysfunction
* Parents who are unable to give informed consent

Ages: 22 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gene expression via Illumina RNA sequencing | Day 3 and 10 post-surgery
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3 and 10 in arginine deficient postoperative infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those involved in T-cell function and associated inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.

SECONDARY OUTCOMES:
Gene expression via Illumina RNA sequencing | Days 3, 10 and 30 post-surgery
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient postoperative infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those involved in T-cell function and associated inflammatory pathways. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
  Secondary analysis will include Day 30 measurements.
Gene expression via Illumina RNA sequencing | Days 3, 10 and 30 post-surgery
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient postoperative infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those known to be associated with necrotising enterocolitis (NEC). Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
Gene expression via Illumina RNA sequencing | Days 3, 10 and 30 post-surgery
  RNA will be extracted from whole blood and sent for Illumina RNA sequencing. These sequences are then mapped to reference gene sets for gene expression analysis. The pattern of alteration in gene expression between days 3, 10 and 30 in arginine deficient postoperative infants after correction of their deficiency by supplementation with arginine will be analysed. The changes in gene expression will be compared with those seen in unsupplemented infants. The genes of interest are those known to be involved with arginine metabolism. Statistical pathway analysis will be used to identify these genes and their relationship with key biological pathways.
Blood ammonia levels | Days 3, 10 and 30 post-surgery
  Blood ammonia levels will be measured at day 3, 10 and 30 post-surgery and levels in supplemented intervention infants will be compared to unsupplemented control infants.
Plasma arginine levels | Days 3, 10 and 30 post-surgery
  Plasma arginine levels will be measured at day 3, 10 and 30 post-surgery and levels in supplemented intervention infants will be compared to unsupplemented control infants.
Plasma proline levels | Days 3, 10 and 30 post-surgery
  Proline is a urea cycle intermediate involved in arginine metabolism. Plasma proline levels will be measured at day 3, 10 and 30 post-surgery. Metabolomics profiling and analysis will be used to compare supplemented intervention infants with unsupplemented control infants.
Body composition measuring total body fluid measured in litres | Days 3, 10 and 30 post-surgery
  Body composition measurements will be taken regularly via bioelectrical impedance measuring total body fluid (intracellular and extra cellular distribution) during the study period. Results from control and intervention infants will be compared.
Body composition measuring fat free mass in grams | Days 3, 10 and 30 post-surgery
  Body composition measurements will be taken regularly via bioelectrical impedance measuring fat free mass during the study period. Results from control and intervention infants will be compared.
Growth measuring body weight in grams | Days 3, 10 and 30 post-surgery
  Infants will be weighed regularly during the study period. Measurements from control and intervention infants will be compared.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Alder Hey Children's Hospital, Liverpool, Merseyside
  - Liverpool Women's Hospital, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available.